CLINICAL TRIAL: NCT03255590
Title: Training and Non-Invasive Brain Stimulation in Chronic Stroke Reduce Abnormal Hand Synergy
Brief Title: Can we Train Patients With Chronic Stroke Out of Abnormal Hand Synergy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NA_00082367; 2R01HD053793-09A1 (NIH)
Record Dates: First submitted 2017-05-18; First posted 2017-08-21 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Cerebral Stroke
Keywords: motor recovery; motor learning; ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Finger Dexterity Training (Experimental): Chronic stroke patients (i.e. great than 6 months) with ischemic stroke confirmed by CT or MRI, residual unilateral upper extremity weakness, able to give informed consent, and able to understand the tasks involved.
  Participants trained for 5 consecutive days, 3 to 4 h/d, on a multi-finger piano-chord-like task that cannot be performed by compensatory actions of other body parts (e.g., arm). Participants had to learn to simultaneously coordinate and synchronize multiple fingers to break unwanted flexor synergies.
  Interventions: Behavioral: Configuration task

INTERVENTIONS:
Behavioral: Configuration task — Training the impaired hand on a configuration task

SUMMARY:
This study plans to determine whether training can change abnormal flexion synergy in chronic stroke patients.

DETAILED DESCRIPTION:
The aim of the current study is to investigate whether motor training in chronic stroke patients can change their abnormal flexion synergy. The investigators will study chronic stroke patients , who are defined as patients that sustained a stroke at least 6 months prior to our testing date.

Three functional aspects of each finger will be tested: maximal voluntary contraction (MVC), finger dexterity, and hand posture.

Prior to intervention, participants will have a baseline assessment including clinical tests, MVC, the individuation task, and the configuration task. Following the baseline assessment patients will receive intervention, training on the configuration task for 5 consecutive days. On the sixth day and as a one week follow-up after, subjects will have a post-intervention assessment containing the same tests performed in baseline.

This design will allow us to determine speed and accuracy during the configuration task, the individuation index, and possible changes in abnormal flexion synergy.

We initially registered the study as two arms (anodal tDCS and sham tDCS groups) but decided to make it one arm due to the number of participants we were able to recruit.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 and older
* Ischemic stroke greater than six months ago, confirmed by CT or MRI
* Residuals unilateral upper extremity weakness
* Ability to give informed consent and understand the tasks involved.
* Appearance of Flexion synergy in hand.
* Ability to extent finger at least for 5 degrees.

Exclusion Criteria:

* Cognitive impairment, with score on Montreal Cognitive assessment (MoCA) ≤ 20
* History of physical or neurological condition that interferes with study procedures or assessment of motor function (e.g. severe arthritis, severe neuropathy, Parkinson's disease)
* Contraindication to tDCS (deep brain stimulators or other metal in the head, skull defect, pacemaker)
* Inability to sit in a chair and perform upper limb exercises for one hour at a time
* Participation in another upper extremity rehabilitative therapy study or tDCS study during the study period
* Terminal illness
* Social and/or personal circumstances that interfere with ability to return for therapy sessions and follow up assessments
* Pregnancy
* Severe Neglect

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Individuation Index | Change from Baseline Individuation Index at 2 weeks
  The relationship between forces (in Newton) in active vs passive fingers during a set of isolated finger movements. It is a measure of finger independence.
Action Research Arm Test (ARAT) | Change from Baseline ARAT at 2 weeks
  Assesses upper limb functioning in activities of daily living using observational methods. It is a 19 item measure divided into a 4-point ordinal scale ranging from:
  3: Performs test normally 2: Completes test, but takes abnormally long or has great difficulty
  1: Performs test partially 0: Can perform no part of test.
  Possible score range of 0 to 57; higher scores equal less impairment.
Fugl-Meyer (Motor Function - Upper Extremity Subscale) | Change from Baseline Impairment Index at 2 weeks
  Assesses functional mobility using observational methods. It is a 66 item measure. Its items are scored on a 3-point ordinal scale.
  0: Cannot perform
  1. performs partially
  2. performs fully
  Possible score range from 0 - 66
Accuracy (Euclidian norm) | Change from Baseline Accuracy at 2 weeks
  The deviation of each finger from a target amount of force generation during a set of finger movements.

SECONDARY OUTCOMES:
Execution Time | Change from Baseline Execution Time at 2 weeks
  The time period from cue appearance to the first moment when finger forces reach the required target. Lower values equal faster execution time.
Semmes Weinstein Monofilament Examination (SWME) | Change from Baseline SWME at 2 weeks
  A quantitative method to systematically assess the threshold stimulus necessary for perception of light touch to deep pressure by using monofilaments of different sizes.
  Interpretation scale for monofilaments:
  2.83 Normal 3.61 Diminished light touch 4.31 Diminished protective sensation 4.56 Loss of protective sensation 6.65 Deep pressure sensation only
Modified Ashworth scale | Change from Baseline Modified Ashworth Scale at 2 weeks
  Tests resistance to passive movement about a joint with varying degrees of velocity in order to assess muscle spasticity.
  Scoring:
  0 No increase in muscle tone
  1 Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension.
  1+ Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the Range of motion (ROM).
  2 More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved.
  3 Considerable increase in muscle tone, passive movement difficult.
  4 Affected part(s) rigid in flexion or extension

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Celnik, Principal Investigator — Department of Physical Medicine and Rehabilitation Johns Hopkins University
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No